CLINICAL TRIAL: NCT04624919
Title: Comparison of Fatigue in Varying Hot Environments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Primary Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00004012
Record Dates: First submitted 2020-10-30; First posted 2020-11-12 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: Randomized, counterbalanced crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot/Dry (Active Comparator)
  Interventions: Other: Hot/Dry
- Warm/Humid (Experimental)
  Interventions: Other: Warm/Humid

INTERVENTIONS:
Other: Hot/Dry — Work is completed in a hot/dry environment.
  Arms: Hot/Dry
Other: Warm/Humid — Work is completed in a warm/humid environment
  Arms: Warm/Humid

SUMMARY:
The purpose of this study is to determine the impact of varying hot environments on physiological and perceptual fatigue during work.

DETAILED DESCRIPTION:
After providing written informed consent and screening, subjects will complete two experimental visits during which they will complete treadmill work in either a hot/dry or warm/humid environment.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 y old men and women
* Self-reported to be healthy

Exclusion Criteria:

* History of any cardiovascular, neurologic, renal, or metabolic disease
* Current tobacco use or regular use within the last 2 years
* Current musculoskeletal injury
* Taking medications with known thermoregulatory or cardiovascular effects (e.g., aspirin, acetaminophen, ibuprofen, beta blockers, diuretics, psychotropics, etc.)
* Currently pregnant or breastfeeding, or planning to become pregnant during the study
* Inability to follow the rules of the protocols or understand the consent form
* Contraindications of consuming a core temperature monitoring pill

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Smoothness of movement | 90 minutes
  The variable, jerk, determines smoothness or unevenness of physical movement during work. This is measured using accelerometers placed along the spine, ankle, and shoulder.
Energy Expenditure | 90 minutes
  The amount of energy the body is expending during work. This is measured using indirect calorimetry.

SECONDARY OUTCOMES:
Perceptual fatigue | 90 minutes
  The degree of fatigue that the subjects perceive during work. This is measured using a subjective likert 0-10 scale named the Fatigue Scale with 0 indicting "no fatigue at all" and 10 indicating "completely fatigued".

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research and Exercise in Special Environments, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data can be made available upon written request.

REFERENCES:
- [Derived] Bartman NE, Vargas NT, Cavuoto LA, Hostler D, Pryor RR. Heat strain differences walking in hot-dry and warm-wet environments of equivalent wet bulb globe temperature. Temperature (Austin). 2024 Aug 26;11(4):333-349. doi: 10.1080/23328940.2024.2384185. eCollection 2024. PMID 39583902